CLINICAL TRIAL: NCT04521270
Title: Financial Burden Associated With Stroke Rehabilitation
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/Lhr/20/2028 Rimsha Tariq
Record Dates: First submitted 2020-08-18; First posted 2020-08-20 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Stroke
Keywords: Financial Burden; Stroke; Longitudinal
MeSH Terms: conditions — Stroke; Financial Stress

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Stroke is one of the main causes of disability and the fourth leading cause of death. All over the world, stroke prevalence varies between 1.9% and 4.3%among adults older than 20 years. The incidence of a stroke increases rapidly with age, double every decade after 55 years old. After a stroke, survivors may experience several issues (i.e. rehabilitation) that increase their direct costs. Stroke survivors and their families may face considerable stroke-related financial burden. To evaluate the total amount or costs use for formal and informal care and the equipment or materials needed for care. This study will be conducted to evaluate the Financial Burden associated with stroke Survivors rehabilitation during their first post stroke year and to analyze the basic predictors of these financial expenses. Data will be collected from Sheikh Zayed hospital Lahore. A cross sectional Longitudinal study will be conducted. The Study will be conducted within 6 months of time period. Post stroke patients who discharge from hospital, after this disease had directly impacts on the survivors' and their family's lives and requires a long rehabilitation process, so they faces many challenges which will be studied. The Barthel Index Scale and Modified Charlson Co-morbidity Index is used to examine the participants autonomy in everyday life activities and their co-morbidities were administered in Stroke Survivors. Stroke Survivors who willing to participate will join in this study and the signed informed consent form will be taken from all participants. After getting approval from research committee data will be collected from the participants and SPSS V 25 will be used for data entry and analysis. The results of this study will help to explore the total amount of cost which use in stroke survivors rehabilitation process.

DETAILED DESCRIPTION:
Stroke is a clinical syndrome characterized by the rapid onset of focal neurological signs, lasting more than 24 hours or leading to death, with a presumed vascular cause. The main causes of stroke is it occur due to infarction and due to hemorrhage. In the U.S, approximately 40 percent of people who die from stroke are male, with 60 percent of deaths occurring in females. Worldwide, cerebro-vascular accidents (stroke) are the second leading cause of death and the third leading cause of disability. Stroke, the sudden death of some brain cells due to lack of oxygen when the blood flow to the brain is lost by blockage or rupture of an artery to the brain, is also a leading cause of dementia and depression. Globally, 70% of strokes and 87% of both stroke-related deaths and disability-adjusted life years occur in low- and middle-income countries. Over the last four decades, the stroke incidence in low- and middle-income countries has more than doubled. During these decades stroke incidence has declined by 42% in high-income countries.

The incidence of a stroke increases rapidly with age, doubling every decade after 55 years old. There are various risk factors for stroke, including both modifiable (e.g., diet, co-morbid conditions) and non-modifiable risk factors (e.g., age, race).Other risk factors which is short-term risks or triggers (e.g., infectious events, sepsis, stress), intermediate- term risk factors (e.g., hypertension, hyperlipidemia) and long-term risk factors for stroke (e.g., sex, race). Risk factors for stroke in the young also likely differ from those in older patients. Recovery and rehabilitation is the most important aspects of stroke treatment. In most strokes cases the patient recover quickly, and sometimes patient recovery is variable. Rehabilitation process includes physical therapy, speech therapy and occupational therapy. Physical therapy involves using exercise and other physical means (e.g., massage, heat) and may help patients to regain their ROM and use of their arms and legs and prevent muscle stiffness in patients or with permanent paralysis. Speech therapy may help patients regain the ability to speak. Occupational therapy may help patients regain independent function and re-learn basic skills (e.g., Getting dressed, preparing a meal and bathing). Stroke is a common, serious, and disabling global health-care problem, and rehabilitation is a major part of patient care.Potentially beneficial treatment options for motor recovery of the arm include constraint-induced movement therapy and robotics. Most favorable interventions that could be beneficial to improve aspects of gait include fitness training, high-intensity therapy, and repetitive-task training.

ELIGIBILITY:
Inclusion Criteria:

* Stroke diagnosed by computerized axial tomography or a magnetic resonance imaging scan.
* Willing to give Informed consent
* Discharged from a rehabilitation hospital

Exclusion Criteria:

* Pre existing Physical or Psychiatric disabilities ( e.g. , Dementia, Multiple Sclerosis, Parkinson's Disease)
* Previous Stroke or Aphasia
* A patient with Reduced level of Consciousness

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were hospitalised within 72 hours of the onset of a first-ever stroke (ischaemic or haemorrhagic), as defined by the World Health Organization (WHO) underwent outpatient rehabilitation in UMMC, and had a caregiver were eligible for inclusion in the present study. Patients were excluded from the study if they were pre-morbidly dependent and/or had subarachnoid haemorrhage, transient ischaemic attack, epilepsy, psychiatric illness or any terminal illness that could affect their daily function and activities.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Structured Questionnaire | 6 Months
  A questionnaire that consisted of three sections:
  1. the patient's sociodemographic data (i.e. age, gender, ethnicity, marital status, employment status, education level and income level), and the caregiver's job, education level and income level;
  2. stroke characteristics, including type of stroke (i.e. ischaemic or haemorrhagic), severity of stroke (measured using the National Institute of Health Stroke Scale [NIHSS]), length of hospital stay and stroke risk factors
  3. stroke-related costs incurred by the patients. The family members of the patients were interviewed three times within the first three months following stroke, and the costs were averaged for analysis.

SECONDARY OUTCOMES:
Modified Charlson Co-morbidity Index | 6 Months
  The use of comorbidities for prognostic assessment has been extensively studied in other fields of medicine. One of the most commonly used comorbidity models is the Charlson Comorbidity Index (CCI), which is based on comorbid conditions with varying assigned weights, resulting in a composite score.
Barthel Index (BI) | 6 Months
  The Barthel Scale/Index (BI) is an ordinal scale used to measure performance in activities of daily living (ADL). Ten variables describing ADL and mobility are scored, a higher number being a reflection of greater ability to function independently following hospital discharge.Time taken and physical assistance required to perform each item are used in determining the assigned value of each item. The Barthel Index measures the degree of assistance required by an individual on 10 items of mobility and self care ADL

CONTACTS AND LOCATIONS:
Overall Officials: Danish Hassan, PhD*, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Riphah International University, Lahore, Punjab Province
  - Riphah Rehabiliation Clinic, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feigin VL, Krishnamurthi RV, Parmar P, Norrving B, Mensah GA, Bennett DA, Barker-Collo S, Moran AE, Sacco RL, Truelsen T, Davis S, Pandian JD, Naghavi M, Forouzanfar MH, Nguyen G, Johnson CO, Vos T, Meretoja A, Murray CJ, Roth GA; GBD 2013 Writing Group; GBD 2013 Stroke Panel Experts Group. Update on the Global Burden of Ischemic and Hemorrhagic Stroke in 1990-2013: The GBD 2013 Study. Neuroepidemiology. 2015;45(3):161-76. doi: 10.1159/000441085. Epub 2015 Oct 28. PMID 26505981
- [Background] Luengo-Fernandez R, Paul NL, Gray AM, Pendlebury ST, Bull LM, Welch SJ, Cuthbertson FC, Rothwell PM; Oxford Vascular Study. Population-based study of disability and institutionalization after transient ischemic attack and stroke: 10-year results of the Oxford Vascular Study. Stroke. 2013 Oct;44(10):2854-61. doi: 10.1161/STROKEAHA.113.001584. Epub 2013 Aug 6. PMID 23920019
- [Background] Luengo-Fernandez R, Gray AM, Rothwell PM; Oxford Vascular Study. A population-based study of hospital care costs during 5 years after transient ischemic attack and stroke. Stroke. 2012 Dec;43(12):3343-51. doi: 10.1161/STROKEAHA.112.667204. Epub 2012 Nov 15. PMID 23160884
- [Background] Tyagi S, Koh GC, Nan L, Tan KB, Hoenig H, Matchar DB, Yoong J, Finkelstein EA, Lee KE, Venketasubramanian N, Menon E, Chan KM, De Silva DA, Yap P, Tan BY, Chew E, Young SH, Ng YS, Tu TM, Ang YH, Kong KH, Singh R, Merchant RA, Chang HM, Yeo TT, Ning C, Cheong A, Ng YL, Tan CS. Healthcare utilization and cost trajectories post-stroke: role of caregiver and stroke factors. BMC Health Serv Res. 2018 Nov 22;18(1):881. doi: 10.1186/s12913-018-3696-3. PMID 30466417
- [Background] Luengo-Fernandez R, Yiin GS, Gray AM, Rothwell PM. Population-based study of acute- and long-term care costs after stroke in patients with AF. Int J Stroke. 2013 Jul;8(5):308-14. doi: 10.1111/j.1747-4949.2012.00812.x. Epub 2012 May 9. PMID 22568484